CLINICAL TRIAL: NCT01459757
Title: A Non-Interventional Retrospective Correlation Of Tumor Mutation Status To Clinical Benefit From The SU011248, A6181036 Treatment Protocol Titled: A Treatment Protocol For Patients With Gastrointestinal Stromal Tumor Who Are Ineligible For Participation In Other SU011248 Protocols And Are Refractory To Or Intolerant Of Imatinib Mesylate
Brief Title: Non-Interventional Retrospective Correlation Of Tumor Mutational Status To Clinical Benefit Of GIST Patients Treated With Sunitinib
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181199
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: GIST
Keywords: Retrospective; GIST; sunitinib; mutational

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Data generated from the past sunitinib A6181036 GIST study
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — Non-interventional; Mutational status data analyzed previously but not collected in the A6181036 study, will be correlated wth A6181036 clinical outcomes data collected during the A6181036 study.

SUMMARY:
Retrospective correlation of clinical outcomes data with mutational status in GIST subjects treated with sunitinib.

DETAILED DESCRIPTION:
This is a non-interventional trial. No active patients will participate in this study. Only data generated from the A6181036 study will be utilized for correlational purposes. The A6181036 study data in addition to mutational status data previously analyzed but not collected as part of the A6181036 study in the same patient population

ELIGIBILITY:
Inclusion Criteria:

* GIST subjects that participated in the A6181036 study that had mutational status data analyzed.

Exclusion Criteria:

* Subjects not participating in the A6181036 study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical outcomes data generated from the sunitinib A6181036 study in GIST correlated with mutational status data previously analyzed for the same patients but not collected as part of the A6181036 study.
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2011-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Mutational status data retrospectively accessed correlated with A6181036 clinical outcomes data in GIST subjects treated with sunitinib | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (36):
- United States (12):
  - City of Hope, Duarte, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Davis Cancer Pavilion and Shands Medical Plaza, Gainesville, Florida
  - Shands Cancer Hospital at the University of Florida, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Masonic Cancer Center - Clinical Trials Office, Minneapolis, Minnesota
  - Oregon Health and Science University, Portland, Oregon
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington, Seattle, Washington
- Australia (3):
  - Prince of Wales Hospital, Oncology Day Center, Randwick, New South Wales
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Peter MacCallum Cancer Institute, Department of Medical Oncology, East Melbourne, Victoria
- UZ Leuven, Leuven, Belgium
- Hopital Notre-dame du Centre Hospitalier Universitaire de Montreal, Montreal, Quebec, Canada
- Herlev Hospital, Herlev, Denmark
- Helsingin yliopistollinen keskussairaala/Syopatautien klinikka, Helsinki, Finland
- France (3):
  - Institut Bergonie, Bordeaux, France
  - CHU La Timone, Service d'Oncologie Medicale, Marseille, France
  - Centre L� B�rd, Lyon, Lyon Cedex
- Germany (3):
  - HELIOS Klinikum Berlin-Buch, Klinik fuer Interdisziplinaere Onkologie, Berlin
  - Klinikum der Universitaet zu Koeln, Cologne
  - Schwerpunktpraxis fuer ambulante Tumortherapie, Düsseldorf
- Tata Memorial Centre, Mumbai, Maharashtra, India
- Leids Universitair Medisch Centrum/ Klinische Oncologie, Leiden, Netherlands, Netherlands
- Klinika Nowotworow Tkanek Miekkich i Kosci, Warsaw, Poland, Poland
- Narodny Onkologicky ustav, Bratislava, Slovakia
- South Korea (2):
  - Seoul National University Hospital/Department of Internal Medicine, Seoul
  - Asan Medical Center, Department of Internal Medicine, Seoul
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
- Centre Hospitalier Universitaire Vaudois, Lausanne, Lausanne, Switzerland
- United Kingdom (2):
  - Sarcoma Unit, London
  - Christie Hospital NHS Trust, Manchester

REFERENCES:
- [Derived] Reichardt P, Demetri GD, Gelderblom H, Rutkowski P, Im SA, Gupta S, Kang YK, Schoffski P, Schuette J, Soulieres D, Blay JY, Goldstein D, Fly K, Huang X, Corsaro M, Lechuga MJ, Martini JF, Heinrich MC. Correlation of KIT and PDGFRA mutational status with clinical benefit in patients with gastrointestinal stromal tumor treated with sunitinib in a worldwide treatment-use trial. BMC Cancer. 2016 Jan 15;16:22. doi: 10.1186/s12885-016-2051-5. PMID 26772734
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181199&StudyName=Non-Interventional%20Retrospective%20Correlation%20Of%20Tumor%20Mutational%20Status%20To%20Clinical%20Benefit%20Of%20GIST%20Patients%20Treated%20With%20Sunitinib